CLINICAL TRIAL: NCT06041113
Title: Recurrent Extrahepatic Bile Duct Stones as a Late Complication of ERCP in Patients With Coexisting Intra- and Extrahepatic Bile Duct Stones：a Long-term Retrospective Cohort Study
Brief Title: Recurrent Extrahepatic Bile Duct Stones as a Late Complication of ERCP in Patients With Coexisting Intra- and Extrahepatic Bile Duct Stones
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Other Study IDs: KY20232281-C-1
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Intrahepatic Bile Duct Stone; Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of coexisting intrahepatic bile duct (IBD) and extrahepatic bile duct (EBD) stones is complicated and requires a multidisciplinary approach. The long-term clinical outcomes of patients initially treated with endoscopic retrograde cholangiopancreatography (ERCP) EBD stone extraction remain unclear. Investigators conducted a retrospective study of patients with coexisting IBD and EBD to investigate the long-term impact of ERCP on the incidence of recurrent EBD stones and to identify risk factors of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* non-gastrointestinal tract reconstruction patients with coexisting IBD and EBD stones who underwent ERCP between July 2008 and December 2020 at Xijing Hospital in China

Exclusion Criteria:

* patients with benign or malignant EBD strictures
* sclerosing cholangitis
* suspected choledochal cysts
* liver cirrhosis
* parasitic liver diseases
* long-term biliary drainage with biliary stents or percutaneous tubes
* without a definitive IBD stone or with a diagnosis of liver calcification as determined by imaging review
* medical records or follow-up information was unavailable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with intrahepatic and extrahepatic bile duct stones who underwent ERCP choledocholithotomy were eligible for our study
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of EBD stones | up to 2 years
  Stone recurrence was defined as new EBD stone formation beyond 3 months after complete initial clearance.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Result] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521